CLINICAL TRIAL: NCT01788592
Title: Prospective Evaluation of Drug-Eluting Stents in Routine Clinical Practice
Brief Title: Prospective Evaluation of Drug-Eluting Stents in Routine Clinical Practice (ASAN PCI Registry)
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2013-02
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Drug eluting stent: Patients who receiving drug eluting stents

SUMMARY:
The objective of this study is to evaluate effectiveness and safety of drug-eluting stent implantation in the "real world" daily practice.

ELIGIBILITY:
Inclusion Criteria:

* coronary disease amenable to percutaneous coronary intervention (PCI)
* no clinical and lesion limitations

Exclusion Criteria:

* patients with a mixture of several drug eluting stents
* terminal illness with life expectancy less than 1 year
* patients with cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients amenable to percutaneous coronary intervention with drug eluting stents
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2003-01 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Event | 1year
  Death from any causes, myocardial infarction or any repeat revascularization

SECONDARY OUTCOMES:
all cause Death | 1year
Myocardial Infarction | 1year
The composite of Death or myocardial infarction | 1year
Any repeat revascularization | 1year
Target vessel revascularization | 1year
Target lesion revascularization | 1year
New lesion revascularization | 1year
Stent thrombosis by Academic Research Consortium criteria | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Park SJ, Ahn JM, Park GM, Cho YR, Lee JY, Kim WJ, Han S, Kang SJ, Park DW, Lee SW, Kim YH, Lee CW, Mintz GS, Park SW. Trends in the outcomes of percutaneous coronary intervention with the routine incorporation of fractional flow reserve in real practice. Eur Heart J. 2013 Nov;34(43):3353-61. doi: 10.1093/eurheartj/eht404. Epub 2013 Oct 2. PMID 24092248